CLINICAL TRIAL: NCT06257953
Title: The Effects of Body Mass Index on Erector Spina Plane Block Analgesia Treatment in Lumbar Disc Herniation Surgery
Brief Title: The Effects of Body Mass Index on Erector Spinae Plane Block Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-BADEK-2024-035
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pain; Pain Postoperative; Pain Acute; Erector Spinae Plane Block; Lumbar Disc Herniation; Body Mass Index
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with a BMI of 18-24.9 kg/m2 (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 15 ml of 0.25% bupivacaine was injected into the area. Then the block process will be applied to the other side in the same way. A total of 30 ml of 15 ml 0.25% bupivacaine will be injected.
  Interventions: Procedure: Erector spinae plane block
- Patients with a BMI of 25-29.9 kg/m2 (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 15 ml of 0.25% bupivacaine was injected into the area. Then the block process will be applied to the other side in the same way. A total of 30 ml of 15 ml 0.25% bupivacaine will be injected.
  Interventions: Procedure: Erector spinae plane block
- Patients with a BMI of 30-40 kg/m2 (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 15 ml of 0.25% bupivacaine was injected into the area. Then the block process will be applied to the other side in the same way. A total of 30 ml of 15 ml 0.25% bupivacaine will be injected.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Erector spinae plane block will be applied to the patients under real-time ultrasound guidance.

SUMMARY:
In recent years, obesity has become one of the leading health problems worldwide. It is known that obesity can cause various diseases and negatively impact the quality of life. Therefore, many conditions believed to be affected by obesity and relevant to patients' quality of life have been scientifically investigated and continue to be researched. One of these conditions is postoperative pain, with studies in the literature indicating that postoperative pain levels increase in parallel with each unit increase in BMI.

The incidence of lumbar disc herniation (LDH) is on the rise and adversely affecting the quality of life. The primary surgical intervention for LDH is discectomy. In recent years, various less invasive techniques, such as microdiscectomy, have been described to improve both surgical and analgesic outcomes. However, even with microdiscectomy surgery, postoperative pain may occur, and its control should be well-managed. Inadequate pain control can lead to unwanted effects of postoperative pain. Regional analgesia techniques may be preferred for effective analgesic treatment after spinal surgery. Methods such as paravertebral block, erector spinae plane block (ESPB), thoracolumbar interfascial plane block are widely used for analgesia in spinal surgery. The effectiveness of these regional techniques may vary depending on various factors, one of which is BMI.

The hypothesis in this study is that as BMI increases, the level of pain in patients may also increase. As a result, this study aims to investigate the relationship between BMI and postoperative pain levels in patients undergoing standard LDH surgery, anesthesia, and analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA physical status I-II-III
* BMI 18 to 40 kg/m2
* Elective LDH surgery

Exclusion Criteria:

* Patient refusing the procedure
* Patients who have previously undergone spinal surgery
* Chronic opioid or analgesic use
* Patients who will operate under emergency conditions
* Patients who will not undergo LDH surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 1st hour after surgery.
  Pain will be assessed at the first-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 1st hour after surgery.

SECONDARY OUTCOMES:
Pain Scores | 2nd hour after surgery.
  Pain will be assessed at the 2nd-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 6th hour after surgery.
  Pain will be assessed at the 6th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 12th hour after surgery.
  Pain will be assessed at the 12th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 24th hour after surgery.
  Pain will be assessed at the 24th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Intraoperative remifentanil consumption | During the intraoperative period
  The amount of remifentanil that patients need to maintain anesthesia during the intraoperative period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)